CLINICAL TRIAL: NCT06588569
Title: Construction of a Multi-mode Ablation Treatment System and Molecular Imaging Multi-omics Study for Malignant Liver Tumors of Digestive System Origin
Brief Title: Multi-mode Ablation and Molecular Imaging Multi-omics Study for Digestive-Origin Malignant Liver Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Wen-Tao Li, Director of Interventional Therapy Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR20210728
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Liver Cancer; Colorectal Cancer Liver Metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-mode Ablation (Experimental): This arm includes patients with primary liver cancer or colorectal cancer liver metastasis (five cases each, totaling ten cases) who will receive multi-mode ablation, a novel ablation therapy that combines cryoablation and radiofrequency ablation.
  Interventions: Device: Multi-mode tumor treatment system
- Conventional Radiofrequency Ablation (Active Comparator): This arm includes patients with primary liver cancer or colorectal cancer liver metastasis (five cases each, totaling ten cases) who will receive conventional radiofrequency ablation treatment.
  Interventions: Device: Radiofrequency ablation therapeutic apparatus

INTERVENTIONS:
Device: Multi-mode tumor treatment system — The intervention for this arm involves the use of a novel multi-mode tumor treatment system, developed by Shanghai MAaGI Medical Technology Co., Ltd. The system combines cryoablation and radiofrequency ablation in a single device. During the treatment, the tumor tissue is rapidly frozen to create an ice ball larger than the lesion by 5mm, followed by thawing and rewarming. Subsequently, the lesion is treated with radiofrequency ablation according to conventional procedures to ensure complete ablation within a safety margin of 5-10mm around the tumor.
  Other Names: MTT-P1
  Arms: Multi-mode Ablation
Device: Radiofrequency ablation therapeutic apparatus — The intervention for this arm involves the use of conventional radiofrequency ablation equipment, which is developed by MedSphere International (Shanghai) Co., Ltd.. During the treatment, the tumor is ablated using predefined power and time settings to ensure complete ablation within a safety margin of 5-10mm around the tumor.
  Other Names: S-1500
  Arms: Conventional Radiofrequency Ablation

SUMMARY:
This single-center, parallel-controlled clinical trial aims to establish a multi-mode ablation system for liver malignant tumors originating from the digestive system. The study will evaluate the safety and efficacy of multi-mode tumor ablation, utilizing a multi-mode imaging platform for ablation planning and immediate evaluation of intraoperative ablation effects. Additionally, the study will employ multi-omics and multi-mode imaging techniques to explore the spatiotemporal heterogeneity and immune escape mechanisms of liver metastases from gastrointestinal tumors, providing guidance for treatment strategy formulation and prognostic evaluation.

DETAILED DESCRIPTION:
This is a single-center, parallel-controlled clinical trial. The study includes a total enrollment of 20 subjects. 10 patients with primary liver cancer will be divided into an experimental group and a control group (5 cases per group); 10 patients with Colorectal Cancer Liver Metastases will also be divided into the experimental group and the control group (5 cases per group). The purpose is to validate the safety and efficacy of multi-mode tumor ablation for liver malignant tumors, aiming to establish a multi-mode tumor treatment system and obtain multi-dimensional biomedical information from patients before, during and after ablation.

The study will employ an interdisciplinary approach, integrating statistics, machine learning and artificial intelligence, to establish a new technical system for rapid efficacy evaluation. Additionally, it will establish a multi-omics artificial intelligence-assisted diagnostic and evaluation system based on radiomics. The system will use artificial intelligence algorithms to automatically locate and identify lesions based on imaging guidance information and accurately predict individual prognoses and anti-tumor immune states through comprehensive preoperative, intraoperative, and postoperative evaluations, providing an important basis for treatment planning, intraoperative dose adjustment, and subsequent treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and 75 years, gender not specified;
2. Pathologically confirmed primary liver cancer or colorectal cancer liver metastases, which is unresectable, intolerant to surgical resection, or refused surgical resection;
3. Intrahepatic lesions with a diameter of ≤4cm, and the number of lesions ≤3.;
4. At least 3 months since the last systemic treatment and at least 1 month since the last local treatment;
5. Child-Pugh class A or B;
6. ECOG PS ≤ 2.

Exclusion Criteria:

1. Liver function Child-Pugh class C , severe jaundice, especially obstructive jaundice;
2. Diffuse liver cancer, or with tumor thrombi in the main portal vein to secondary branches or hepatic vein;
3. Significant liver atrophy, tumor volume too large, requiring ablation range of up to one-third of the liver volume;
4. Multiple systemic metastases, expected survival < 3 months;
5. Recent history of esophageal (gastric fundus) variceal bleeding within the past month;
6. Severe functional failure of major organs such as the liver, kidneys, heart, lungs or brain;
7. Presence of active infection;
8. Uncorrectable coagulation dysfunction and severe hematological abnormalities, with a significant bleeding tendency;
9. Refractory massive ascites, pleural effusion, or cachexia;
10. Pregnancy, disorder or inability to cooperate with treatment;
11. Any other factors deemed inappropriate for inclusion or affecting the subject's participation in the study, as determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Antitumor immune response | max 24 months
  Antitumor immune response is a measure that evaluates the efficacy of multi-mode ablation in activating a durable and specific immune response against tumor cells. This outcome will be assessed as follows:
  Flow cytometry to quantify the proportions and absolute numbers of immune cell subsets, including CD4+ T cells, CD8+ T cells, NK cells, B cells and dendritic cells (DCs), as well as the immune suppressive myeloid-derived suppressor cells (MDSCs).
  Cytokine profiling is performed to measure the levels of immune-related cytokines such as interferon-gamma (IFN-γ), interleukin-2 (IL-2), and tumor necrosis factor-alpha (TNF-α).
  Assessment of immune memory phenotypes through the analysis of T cell receptor (TCR) repertoire diversity and clonality.
6-month Disease Control Rate | 6 months
  6-month Disease Control Rate (6-month DCR) refers to the proportion of patients who have a complete response (CR), partial response (PR), or stable disease (SD) at the 6-month follow-up visit.

SECONDARY OUTCOMES:
6-Month Progression-Free Survival | 6 months
  6-month progression-free survival (6-month PFS) refers to the percentage of patients who are alive without tumor progression or metastasis six months after the start of treatment.
1-Year Progression-Free Survival | 1 year
  1-year progression-free survival (1-year PFS) refers to the percentage of patients who are alive without tumor progression or metastasis one year after the start of treatment.
1-Year Overall Survival | 1 year
  1-year overall survival (1-year OS) refers to the percentage of patients who are still alive one year after the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Director of Interventional Therapy Department, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China